CLINICAL TRIAL: NCT06091332
Title: Hemorrhagic Brainstem Cavernous Malformations Treatment With Sirolimus: a Randomized, Placebo-controlled Pilot Trial
Brief Title: Hemorrhagic Brainstem Cavernous Malformations Treatment With Sirolimus: aSingle Centre, Randomized, Placebo-controlled Pilot Trial
Acronym: CALM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhu, Vice director of neurosurgey department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-816
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cavernous Malformations; Intracerebral Hemorrhage; Brainstem Stroke
Keywords: Cavernous Malformations; Brainstem; Rebleeding rate; Sirolimus
MeSH Terms: conditions — Cerebral Hemorrhage; Brain Stem Infarctions | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: According to the study protocol, patients were randomly divided into a normal-dose group, low-dose group, and control group at a ratio of 1:1:1. Additionally, to minimize potential bias, this study employed a double-blind approach.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind design means that throughout the entire study, neither the participating patients nor the investigators are aware of which treatment group the patients are assigned to, in order to minimize potential biases. The blinding level is double-blind, which means that both the patients in the treatment group and those in the control group, as well as the investigators, are unaware of the treatment the patients receive, ensuring objectivity and reliability of the study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-dose sirolimus group (Experimental): Participants will receive oral sirolimus with a target blood concentration of 9-15ng/ml continuously for 12 months.
  Interventions: Drug: Sirolimus
- Low-dose sirolimus group (Experimental): Participants will receive oral sirolimus with a target blood concentration of 3-7ng/ml continuously for 12 months
  Interventions: Drug: Sirolimus
- Placebo control group (Placebo Comparator): Participants will receive oral placebo(starch formulation) for 12 months.
  Interventions: Drug: Starch flake

INTERVENTIONS:
Drug: Sirolimus — Sirolimus is an mTORC1 inhibitor that has received approval from the U.S. Food and Drug Administration (FDA) and has recently been successfully used to treat lymphatic malformations and venous/lymphatic malformations associated with the same PIK3CA GOF mutations.
  Other Names: Rapamycin
  Arms: High-dose sirolimus group; Low-dose sirolimus group
Drug: Starch flake — The placebo is composed of starch material and is formulated at 0.5 grams per tablet.
  Arms: Placebo control group

SUMMARY:
The aim of this pilot phase trial is to assess the safety and tolerability, and estimate the efficacy of sirolimus in reducing the incidence of ICH during high-risk periods for rebleeding, compared to placebo. This pilot trial will inform the design of a future definitive clinical trial on sirolimus treatment for CCM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years, any gender;
2. Patients who have experienced their first symptomatic BSCM ICH within the six months before randomisation;
3. Diagnosed with solitary BSCM through T2, GRE/T2*, or SWI MR imaging;
4. ICH within or around the BSCM confirmed by CT /MR;
5. Capable of signing an informed consent form with the accompaniment and understanding of a guardian.

Exclusion Criteria:

1. Cancer history;
2. Pregnancy or lactation;
3. Sirolimus/starch allergy;
4. Modified Rankin Scale (mRS) score 5, respiratory failure or currently severe bleeding requiring life support treatment;
5. Abnormal liver and/or kidney function (transaminase levels greater than 50, creatinine greater than 110), abnormal white blood cell/platelet counts (white blood cell count below 3.5 or above 9.5 x 109/L or exceeding normal values, platelet count below 100 or above 300);
6. History of previous immunosuppressive therapy;
7. History of prior surgical intervention for CCM ;
8. History of prior cranial radiation therapy ;
9. Familial CCM or people with multiple CCM;
10. Patients with concurrent acute active infections (e.g., severe bacterial, viral, or fungal infections);
11. Uncontrolled diabetes mellitus;
12. Currently participating in another clinical trial;
13. Patient unwilling/unable to undergo MRI.
14. Co-administration of drugs affecting CYP3A4 enzymes (ketoconazole, voriconazole, itraconazole, telithromycin, clarithromycin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to explore the safety of sirolimus in the management of BSCMs. | 24 months
  A serious adverse event is an SAE occurring during any study phase that fullfils one or more of the following criteria:
  i. Results in death, ii. Is life-threatening, iii. Requires inpatient hospitalization or prolongation of existing hospitalization, iv. Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, v. Is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above.
  SAE will be assessed at each follow-up visit (15 days, 2 months, 6 months, 12 months, 18 months, 24 months). During the trial, participants can promptly report potential SAEs to the research team via the telephone. We will establish continuous, real-time communication with patients via the telephone, facilitating round-the-clock reporting of potential endpoints or adverse reactions to the clinical trial investigators.

SECONDARY OUTCOMES:
We will measure the tolerability of sirolimus in the management of BSCMs. | 24 months
  Based on prior clinical experience and reports from sirolimus trials, adverse events (AE) have included oral ulcers, upper respiratory tract infections, headaches, respiratory illnesses, stomatitis, seizures, and fever. Other commonly reported AEs are nausea, vomiting, fatigue, dizziness, diarrhea, and mild allergic reactions such as rash or itching. Minor infections, mild gastrointestinal disturbances, and fluctuations in blood pressure or heart rate have also been observed.
  Unanticipated Adverse Device Effect (UADE): Any serious adverse effect on health or safety or any life-threatening problem or death caused by or associated with sirolimus, if that effect, problem or death was not previously identified in nature, severity or degree of incidence in the investigational plan, or any other unanticipated serious problem associated with sirolimus that related to the rights, safety or welfare of subjects.
We will measure the occurrence of recurrent ICH from the BSCM within 24 months. | 24 months
  a. The primary efficacy outcome will be the occurrence of recurrent ICH from the BSCM within 24 months. ICH is defined as the presence of new focal neurological dysfunction or new headache symptoms, and confirmed by head CT/MR imaging examinations indicating new cerebral haemorrhage attributed to BSCM. If the primary efficacy outcome occurs, surgery will be considered for participants with a second ICH during follow-up. Radiosurgery or conservative treatment may also be considered for patients with a high risk of surgical intervention.
We will measure the efficacy outcomes in MR | 24 months
  A secondary efficacy outcome will be change in magnetic susceptibility using quantitative susceptibility mapping (QSM) MRI34 at 24 months after randomisation. Recent studies have described the feasibility, reliability, and validity of QSM as a biomarker for the effect of drugs on CCM.
We will measure several the quality of life | 24 months
  Quality of Life (mRS score and EuroQOL five dimensions questionnaire (EQ-5D) scale) within 24 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhu, Doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ren AA, Snellings DA, Su YS, Hong CC, Castro M, Tang AT, Detter MR, Hobson N, Girard R, Romanos S, Lightle R, Moore T, Shenkar R, Benavides C, Beaman MM, Muller-Fielitz H, Chen M, Mericko P, Yang J, Sung DC, Lawton MT, Ruppert JM, Schwaninger M, Korbelin J, Potente M, Awad IA, Marchuk DA, Kahn ML. PIK3CA and CCM mutations fuel cavernomas through a cancer-like mechanism. Nature. 2021 Jun;594(7862):271-276. doi: 10.1038/s41586-021-03562-8. Epub 2021 Apr 28. PMID 33910229
- [Background] Flemming KD, Graff-Radford J, Aakre J, Kantarci K, Lanzino G, Brown RD Jr, Mielke MM, Roberts RO, Kremers W, Knopman DS, Petersen RC, Jack CR Jr. Population-Based Prevalence of Cerebral Cavernous Malformations in Older Adults: Mayo Clinic Study of Aging. JAMA Neurol. 2017 Jul 1;74(7):801-805. doi: 10.1001/jamaneurol.2017.0439. PMID 28492932
- [Background] Ren J, Huang Y, Ren Y, Tu T, Qiu B, Ai D, Bi Z, Bai X, Li F, Li JL, Chen XJ, Feng Z, Guo Z, Lei J, Tian A, Cui Z, Lindner V, Adams RH, Wang Y, Zhao F, Korbelin J, Sun W, Wang Y, Zhang H, Hong T, Ge WP. Somatic variants of MAP3K3 are sufficient to cause cerebral and spinal cord cavernous malformations. Brain. 2023 Sep 1;146(9):3634-3647. doi: 10.1093/brain/awad104. PMID 36995941